CLINICAL TRIAL: NCT01149629
Title: A Randomized, Open-Label, Three-Period, Three-Sequence, Single-Dose Crossover and Separate Three-Daily-Dose Treatment Period Study Comparing the Pharmacokinetic Profiles Following Oral Dosing of 300 mg of Droxidopa in the Fed Versus Fasted State, the Bioequivalence of Three 100 mg Capsules of Droxidopa Versus a Single 300 mg Capsule of Droxidopa, and 300 mg of Droxidopa Given Three Times at Four Hour Intervals in Healthy, Elderly Subjects
Brief Title: Study of the Fed-Fast Pharmocokinetics and Bioequivalance of 300mg Capsules of Droxidopa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Droxidopa NOH101
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension
Keywords: Droxidopa; Randomized; Crossover; Open Label; Bioequivalence; Fed Fast; TID
MeSH Terms: interventions — Droxidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fed Dosing (Active Comparator): Subjects fed a high calorie, high fat meal prior to receiving 3 x 100mg capsules
  Interventions: Drug: Droxidopa
- Fasted Dosing (Active Comparator): Subjects fasted prior to receiving 3 x 100mg capsules
  Interventions: Drug: Droxidopa
- Bioequivalence (Active Comparator): Subjects fasted prior to receiving 1x 300mg capsule
  Interventions: Drug: Droxidopa
- TID Dosing (Active Comparator): Droxidopa 300 mg given TID
  Interventions: Drug: Droxidopa

INTERVENTIONS:
Drug: Droxidopa — One capsule containing 300 mg droxidopa, given once
  Arms: Bioequivalence
Drug: Droxidopa — 3 capsules each containing 100 mg droxidopa, give 3 times at 4 hour intervals
  Arms: TID Dosing
Drug: Droxidopa — 3 capsules each containing 100 mg droxidopa, given once
  Arms: Fasted Dosing; Fed Dosing

SUMMARY:
One purpose of this study is to determine if taking droxidopa after eating will have an effect on how the body processes (absorbs and eliminates) the drug in healthy elderly subjects. Another purpose of this study is to see how the body processes (absorbs and eliminates) one 300mg capsule compared to three 100mg capsules. This study will also evaluate how well the body processes (absorbs and eliminates) and tolerates droxidopa when a 300 mg capsule is given 3 times a day for a total dose of 900 mg over the course of one day.

Droxidopa is used to treat low blood pressure upon standing in patients with diseases of the nervous system, to prevent low blood pressure in patients with kidney disease during hemodialysis (removal of waste products of the blood), and to treat frozen gait (walking, stepping or running) and dizziness upon standing in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This is a two-part study. Part I is a randomized, open-label, three-period crossover study in 24 healthy, elderly, male or female subjects. Subjects will be allocated to one of three treatment sequences according to a randomization schedule prepared prior to the start of the study. Each subject will receive a single, oral dose of three 100 mg capsules of droxidopa with 240 mL of water either in the fasted state (Treatment A) or immediately following the consumption of a standardized high-fat meal (Treatment B) and a single, oral dose of one 300 mg capsule of droxidopa with 240 mL of water in the fasted state (Treatment C) on Days 1, 4, and 7. Subjects will be discharged from the research clinic on Day 8 after completing all posttreatment follow-up assessments and will return to the research clinic approximately 1 week later for Part II of the study. Part II of the study is an open-label design where all subjects will receive three doses of 300 mg droxidopa (three 100 mg capsules/dose) at 4 hour intervals and will be followed for a concurrent 24 h period.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written consent on an IRB-approved Informed Consent Form (ICF), prior to any study-specific evaluation. Subjects should have the ability to read and understand the ICF, ask for any clarifications from the study staff, and be able to comply with all planned study procedures.
2. Male or female ≥65 years of age.
3. Body mass index (BMI) between 18 and 35 kg/m2, inclusive.
4. If female, not pregnant (or lactating), as evidenced by a negative serum pregnancy test, and is surgically sterile (hysterectomy, bilateral ovariectomy, or bilateral tubal ligation), or at least 2 years postmenopausal.
5. Ability and willingness to abstain from alcohol from 48 h prior to the first dose until the completion of the study.
6. No clinically significant abnormalities on the basis of medical history, physical examination, and vital signs unless currently controlled with medical treatment (e.g., a stable medication dosing regimen).
7. Computerized, 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations, as judged by the investigator.
8. All values for hematology, clinical chemistry, and urinalysis are normal or if abnormal-are deemed not clinically significant as judged by a physician investigator with documented agreement from the Medical Monitor.
9. Nonsmoking or have quit smoking at least 6 months prior to dosing.

Exclusion Criteria:

1. Presence of active or recurring clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease not currently controlled with medical treatment (e.g., a stable medication dosing regimen).
2. Presence of an active malignancy of any type other than nonmelanomatous skin malignancies.
3. History of relevant drug and/or food allergies.
4. Recent history (past 5 years) of alcohol abuse or drug addiction.
5. Required use of concomitant medications that could confound the PK or safety evaluation, such as medications that affect GI function (including proton pump inhibitors or metoclopramide) or vasoconstricting agents (e.g., ephedrine, dihydroergotamine, or midodrine), -triptans (e.g., sumatriptan, naratriptan, zolmitriptan, rizatriptan), halogen-containing anesthetics (e.g., cyclopropane, or halothane), catecholaminecontaining preparations (e.g., isoprenaline), non-selective MAOIs, ergotamine derivatives (except for anti-Parkinson medications), or any drugs with anti-hypertensive properties that in the investigator's opinion, could significantly contribute to the subject's orthostatic hypotension.
6. Participation in an investigational drug study within 30 days prior to study drug administration.
7. Donated a unit of blood (500 mL) or plasma within the 30-day period prior to the initial dose of study medication or who intend to donate blood or plasma within a 30-day period following the final dose of study medication.
8. Positive screen for drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines) or alcohol.
9. Positive screen for urine cotinine.
10. Positive screen for hepatitis B surface antigen.
11. Positive screen for antibodies to hepatitis C virus.
12. Positive screen for antibodies to human immunodeficiency virus (HIV-1/HIV-2).
13. Acute illness within 5 days prior to drug administration.
14. History of coagulation disorder, thrombocytopenia, bleeding tendency, or gastrointestinal bleeding.
15. Professional or ancillary personnel involved in the study.
16. In the opinion of the investigator, not suitable for entry into the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Droxidopa Pharmacokinetics | 24 hours
  Blood samples will be collected at the time from 0 to 24 hours. Cmax, Tmax, AUC(0-∞), AUC(0-t), t1/2, and CL/F, will be determined for plasma concentrations of droxidopa in Parts I and II and will also be determined for two of its metabolites (3-OM-droxidopa and norepinephrine) in Part II only.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Haugen, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Chen JJ, Hewitt LA. Comparison of the Pharmacokinetics of Droxidopa After Dosing in the Fed Versus Fasted State and with 3-Times-Daily Dosing in Healthy Elderly Subjects. Drugs R D. 2018 Mar;18(1):77-86. doi: 10.1007/s40268-018-0226-z. PMID 29392574